CLINICAL TRIAL: NCT05311865
Title: Transmission of Covid-19 During Clubbing Events in Closed Places
Acronym: ITOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Cerballiance (Unknown); Kappa Santé (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ANRS0066s
Record Dates: First submitted 2022-03-08; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Healthy Participant
Keywords: SARS CoV-2; Transmission; vaccinated; Night-club

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, randomized controlled intervention study with 1200 participants distributed 2: 1 in two groups of volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participating to the event (Experimental)
  Interventions: Other: Club event
- Non partipating to the event (No Intervention)

INTERVENTIONS:
Other: Club event — Participate in a club event without a mask, indoors, with vaccinated people.
  Arms: participating to the event

SUMMARY:
The ITOC study is a cluster randomised, controlled, multicentre trial in Paris region, France. The intervention is an 8-hour indoor clubbing event with no mask wearing, no social distancing, at maximum room capacity. 1,200 healthy volunteers aged 18-49 years and fully vaccinated will be included. Participants are recruited by group of up to 10, to be randomized 2:1 to experimental group (800 volunteers in a venue ) or control group (400 volunteers asked to stay at home). All participants will provide a salivary sample the day of experiment and seven days later. Participants will also answer surveys on the social and psychological impact of lockdown and indoor club closing, attitude towards vaccination, behaviour at risk of COVID-19 transmission during the day of the event (for both groups) as well as follow-up surveys on symptoms that participant may experience. Virological analyses include polymerase chain reaction (PCR) of salivary samples and air of the venue, investigating SARS-CoV-2 PCR.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 49 years old
* Vaccination completed
* People who declared to have no risk factor to severe form for Covid-19 disease
* People who declared not to live in the same place as someone with these risk factors
* People residing in Ile-de-France area
* People affiliated with the the French social security citizen scheme

Exclusion criteria:

* Presence of symptoms of COVID in the 2 weeks before the event
* Pregnant woman or woman who declares not having an effective contraception method
* Self identification of medical conditions or comorbidities identified as a proven risk of severe COVID infection
* People living with a person with these risk factors
* Confirmed diagnosis of SARS-CoV-2 within two weeks before the event
* Participants under tutorship or curatorship;
* Underage participants;
* Participants unable to give free and informed consent;
* Participants not affiliated to the French social security citizen scheme: obligation to join a social security scheme or be a beneficiary thereof.
* Participants under legal protection

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1216 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2021-10-17 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
Number of positive RT-PCR at day 7 | Day 7
  Number of participants in each groups with a positive salivary RT-PCR

SECONDARY OUTCOMES:
Number of SARS-CoV-2 infection cases | Day 5 up to day 10
  Numbers of asymptomatic, symptomatic, and severe SARS-CoV-2 infection according to a self-assessment by a questionnaire sent online in each group
Number of participants with seasonal respiratory viruses | Day 0 and day 7
  Number of participants in each group with a positive seasonal respiratory viruses PCR
Number of symptomatic and asymptomatic respiratory infection | Day 5 to day 10
  Numbers of asymptomatic, symptomatic, and severe seasonal respiratory viruses infection according to a self-assessment by a questionnaire sent online
Number of detected virus in the air | Day 0
  Number of detected virus in the air, by the AerosolSense
Number of mutations, deletions and insertions on the viral genome in participants samples | Day 0 and day 7
  Whole genome sequencing of virus detected in participants samples : number of mutations, deletions or insertions on all the viral genes of consensus sequences
Number of mutations, deletions and insertions on the viral genome in Aerosol samples | Day 0 and day 7
  Whole genome sequencing of virus detected in Aerosol samples : number of mutations, deletions or insertions on all the viral genes of consensus sequences
Percentage of divergence between phylogenetic analysis of participants and aerosol samples | Day 0 and day 7
  Establishing the distance matrix between the viruses in participants samples and viruses detected by aerosol sense
Percentage of Health protocol adherence | Day 1
  Percentage of positive responses to a questionnaire assessing degree of adherence to the health protocol by questionnaire sent online to participants and organizers after the evenings.
Percentage of Interactions between the participants during the event | Day 1
  Percentage of responses to a questionnaire assessing number of individual interactions during the event

CONTACTS AND LOCATIONS:
Overall Officials: Yazdan Yazdanpanah, Pr, Study Director — ANRS, Emerging Infectious Diseases
Locations (1):
- ANRS, Paris, France

REFERENCES:
- [Derived] Luong Nguyen LB, Goupil de Bouille J, Menant L, Noret M, Dumas A, Salmona M, Le Goff J, Delaugerre C, Crepey P, Zeggagh J; ITOC Study Group. A Randomized Controlled Trial to Study the Transmission of SARS-CoV-2 and Other Respiratory Viruses During Indoor Clubbing Events (ANRS0066s ITOC Study). Clin Infect Dis. 2023 Dec 15;77(12):1648-1655. doi: 10.1093/cid/ciad603. PMID 37795682
- [Derived] Goupil de Bouille J, Luong Nguyen LB, Crepey P, Garlantezec R, Dore V, Dumas A, Ben Mechlia M, Tattevin P, Gaudart J, Spire B, Lert F, Yazdanpanah Y, Delaugerre C, Noret M, Zeggagh J. Transmission of SARS-CoV-2 during indoor clubbing events: A clustered randomized, controlled, multicentre trial protocol. Front Public Health. 2022 Nov 4;10:981213. doi: 10.3389/fpubh.2022.981213. eCollection 2022. PMID 36438274